CLINICAL TRIAL: NCT04419207
Title: Detecting Lung Cancer by Volatile Organic Compounds in Exhaled Breath: a Study of Lung Cancer Diagnostic Biomarker
Brief Title: Detecting Lung Cancer Based on Exhaled Breath
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Haidian Hospital (Other); Aerospace 731 Hospital (Other); Beijing Breatha Biological Technology Co., Ltd, Beijing (Unknown); The First Affiliated Hospital of Zhengzhou University (Other); Jiangsu Cancer Institute & Hospital (Other)
Responsible Party: Principal Investigator, zhouzuli, M.D.，Department of Thoracic Surgery, Peking University People's Hospital
Other Study IDs: 2019PHB095-01
Record Dates: First submitted 2020-06-04; First posted 2020-06-05 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma; Lung Cancer; NSCLC; Lung Neoplasms
Keywords: volatile organic compounds; exhaled breath; biomarker
MeSH Terms: conditions — Carcinoma; Lung Neoplasms | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled breath samples will be collected with air bags.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Surbery: Patients who with pulmonary nodules in computed tomography and planned to receive thoracic surgery will be included. And those who have other types of cancer, received anti-tumor treatment before surgery, liver disease, or infections will be excluded.
  Interventions: Diagnostic Test: Breath test
- Healthy Controls: Adult participants (>18 yr) who plan to receive annual physical examination and low-dose computed tomography will be included. And those who have history cancers, received anti-tumor treatment before surgery, liver disease, or infections will be excluded.
  Interventions: Diagnostic Test: Breath test

INTERVENTIONS:
Diagnostic Test: Breath test — Exhaled breath of each participant will be collected with air bags and directly detected by a high-resolution high-pressure photon ionization time-of-ﬂight mass spectrometry (HPPI-TOFMS).

SUMMARY:
Early detection is critical to improve the overall survival of lung cancer. Endogenous volatile organic compounds (VOCs) can be derived from many different metabolic pathways. On the other hand, cancer cells have different metabolism patterns compared with normal cells. Thus, detecting VOCs in exhaled breath using highly sensitive mass spectrometry would be a promising approach for lung cancer detection.

DETAILED DESCRIPTION:
Endogenous volatile organic compounds (VOCs) can be derived from many different metabolic pathways. VOCs can be transported to the alveoli through the blood circulation and expelled by exhalation. Changes in VOCs production, clearance, and alterations in lung air-blood exchange functions can lead to aberrant VOCs profiles in the exhaled breath. Testing exhaled breath has the advantages of being completely non-invasive and easy to collect, and has been considered as a perfect approach for disease diagnoses and therapeutic monitoring. Many clinical studies have found that VOCs in exhaled breath are closely related to disease status. Specific VOCs alterations have been identified in many tumors, especially lung cancer.

In this study, we use a highly sensitive mass spectrometry to detect exhaled VOCs of lung cancer patients and healthy people. A lung cancer diagnosis model based on mass spectrometry data and support vector machine will be initially established and validated.

ELIGIBILITY:
Inclusion Criteria for inpatient :

* pulmonary nodules in competed tomography images
* plan to receive thoracic surgery

Inclusion Criteria for controls :

* have planned physical examination every year
* plan to receive low-dose computed tomography

Exclusion Criteria:

* history of malignant tumors.
* receive anti-tumor treatment such as radiotherapy, chemotherapy, targeted therapy before surgery
* with infections or liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible inpatients will be recruited from Department of Thoracic Surgery, Peking University People's Hospital and Beijing Haidian Hospital.
  For healthy controls, eligible participants will be recruited from those who receive planned annual physical examination at Aerospace 731 Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2236 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-01-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity of exhaled breath | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, diagnostic sensitivity of exhaled breath will be calculated
Diagnostic specificity of exhaled breath | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, diagnostic specificity of exhaled breath will be calculated
Positive predictive value of exhaled breath | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, positive predictive value of exhaled breath will be calculated
Negative predictive value of exhaled breath | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, negative predictive value of exhaled breath will be calculated
Diagnostic accuracy of exhaled breath | 2 year
  Using pathologic diagnosis of lung cancer as gold standard, diagnostic accuracy of exhaled breath will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Mantang Qiu, M.D, Study Chair — Peking University People's Hospital Thoracic Surgery Department; Zuli Zhou, M.D, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No